CLINICAL TRIAL: NCT06721442
Title: Effect of Dapagliflozin, a Sodium-Glucose Co-Transporter 2 Inhibitor, on Ventricular Repolarization Electrocardiographic Parameters in Type 2 Diabetes Patients: DAPA - ECG Study
Brief Title: Effect of Dapagliflozin on Electrocardiographic Parameters in Type 2 Diabetes Patients: DAPA - ECG Study
Acronym: DAPA-ECG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Rodrigo Noronha Campos, Doctor-cardiologist, Beneficência Portuguesa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAPA-ECG
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Arrhythmias, Cardiac; Diabetes Mellitus
Keywords: Type 2 Diabetes Cardiac Arrhythmias; Dapagliflozin; Ventricular Repolarization; Electrocardiogram; Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac; Diabetes Mellitus | interventions — dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, open-label, controlled trial
Masking Description: All eligible patients were randomized into two groups using the REDCap software: one group received dapagliflozin combined with optimized medical treatment, while the other group received only the optimized treatment. Each group included 87 patients. To minimize bias in the open-label design, electrocardiograms performed at baseline and at the final visit were evaluated by external independent examiners blinded to group allocation. The Kappa index was used to ensure data consistency and reliability. These measures provided greater rigor and validity to the study results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapafliflozin (Active Comparator): A total of 174 individuals were assessed for eligibility, of whom 87 were randomized to receive dapagliflozin in combination with optimized medical treatment for type 2 diabetes.
  Interventions: Drug: Dapagliflozin (DAPA)
- Control group (No Intervention): A total of 174 individuals were assessed for eligibility, and 87 were randomized to continue receiving optimized medical treatment for type 2 diabetes.

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Patients randomized to receive a daily dose of 10 milligrams of dapagliflozin were evaluated to assess the medication's impact on electrocardiographic parameters of repolarization, with focus on its potential to reduce ventricular repolarization prolongation in individuals with type 2 diabetes.
  Other Names: iSGLT2; SGLT2 inhibitor
  Arms: Dapafliflozin

SUMMARY:
The goal of this clinical trial is to evaluate whether dapagliflozin can reduce ventricular electrical remodeling, as measured by electrocardiographic parameters, in patients with type 2 diabetes (T2D). The study focuses on understanding how dapagliflozin affects the risk of potentially malignant ventricular arrhythmias and sudden cardiac death in this population.

The main questions it aims to answer are:

* Does dapagliflozin reduce the TpTe interval in patients with T2D?
* Does dapagliflozin impact other electrocardiographic parameters such as QT and QTc intervals, TpTe/QT ratio, and QT dispersion?

Researchers will compare patients treated with dapagliflozin plus optimized medical therapy (OMT) o those receiving OMT without SGLT2 inhibitors to assess whether there is a significant difference in the electrocardiographic parameters and ventricular electrical remodeling.

Participants will:

Be randomized into two groups: one treated with dapagliflozin and the other with optimized medical therapy.

Undergo clinical, electrocardiographic, laboratory, and echocardiographic evaluations at baseline and after three months.

This randomized, prospective, multicenter, open-label study seeks to clarify the cardioprotective mechanisms of dapagliflozin, particularly its impact on ventricular electrical remodeling in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Background: In patients with type 2 diabetes (T2D), hyperglycemia and glycemic variability lead to prolongation and greater heterogeneity of ventricular repolarization, manifested on the electrocardiogram through an increase in QT, QTc, TpeakTend (TpTe) intervals and the TpTe/QT ratio, increasing the risk of potentially malignant arrhythmias. Dapagliflozin has demonstrated efficacy in reducing cardiovascular events in diabetic patients at high cardiovascular risk and in the risk of serious ventricular arrhythmias and sudden cardiac death. However, the exact mechanisms by which dapagliflozin confers this protection have not yet been fully elucidated.

Objective: The main objective of the study was to evaluate the impact of dapagliflozin on the TpTe interval of patients with T2D, and secondarily, it examined its impact on various electrocardiographic parameters such as the QT and QTc intervals, the TpTe/QT ratio, QT dispersion, J-T peak interval, QRS-T angle and heart rate.

Methods: This randomized, prospective, multicenter and open-label study involved 174 patients with T2D, divided into two groups: one treated with dapagliflozin and the other with optimized medical therapy without iSGLT2. Clinical, electrocardiographic, laboratory and echocardiographic evaluations were carried out at the beginning and after three months. The statistical analysis included means, standard deviations, quartiles, and frequencies, with 95% confidence intervals, using Chi-square (or Fisher) and t-Test (or Mann-Whitney) for initial differences, and a linear mixed-effects model to evaluate the results, adopting a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old);
* Resting 12-lead electrocardiogram in sinus rhythm;
* Type 2 diabetes;
* Body mass index (BMI), calculated as weight in kilograms divided by height in meters squared, of 45 or less;
* Estimated glomerular filtration rate (eGFR) of at least 30 ml per minute per 1.73 m² of body surface area, according to CKD-EPI criteria;
* Agreed to participate in the study and signed the informed consent form (ICF).

Exclusion Criteria:

* Patients with a QRS interval > 120 ms;
* Insulin use;
* Atrial fibrillation rhythm;
* Cardiac pacemaker rhythm;
* Planned cardiac surgery or angioplasty within 3 months;
* Glycemic control issues (glucose > 240 mg/dL) after an overnight fast of 8 hours in both groups;
* Liver disease, defined by serum levels of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 3 times the upper limit of normal during the baseline phase;
* Medicinal treatment for weight loss within 3 months of the study start;
* Pregnant women, women with delayed menstruation, or those breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Effect of Dapagliflozin on the TpeakTend Interval | 90 days
  In the intervention group (dapagliflozin), 12-lead electrocardiograms (ECGs) were performed during designated outpatient visits, with the initial baseline recording conducted at visit 1 (day 0) and the subsequent recording at the final visit, approximately 90 days after the study began.
  The ECGs were obtained using Micromed electronic equipment, configured with a paper speed of 25 mm/s and an amplitude of 10 mm/mV, ensuring standardized measurements. The ECG intervals were manually measured using Wincardio software (version 11.1.0.0).
  The primary outcome, the interval between the peak of the T wave and the end of the T wave (TpTe), was assessed to evaluate the effect of dapagliflozin. This assessment compared the two time points (baseline and follow-up), with all ECGs analyzed by an independent external examiner to ensure objectivity and reliability of the study results.

SECONDARY OUTCOMES:
Effect of Dapagliflozin on the QT and QTc Interval | 90 days
  In the intervention group (dapagliflozin), 12-lead electrocardiograms (ECGs) were performed during designated outpatient visits, with the initial baseline recording conducted at visit 1 (day 0) and the subsequent recording at the final visit, approximately 90 days after the study began.
  The ECGs were obtained using Micromed electronic equipment, configured with a paper speed of 25 mm/s and an amplitude of 10 mm/mV, ensuring standardized measurements. The ECG intervals were manually measured using Wincardio software (version 11.1.0.0).
  The secondary outcomes, the QT and corrected QT (QTc) intervals, were assessed to evaluate the effect of dapagliflozin. These intervals were analyzed by comparing the two time points (baseline and follow-up). All ECGs were reviewed by an independent external examiner, ensuring objectivity and reliability in the interpretation of the study data.
Effect of Dapagliflozin on the TpTe/QT ratio | 90 days
  To evaluate the effect of dapagliflozin on the TpTe/QT ratio, an electrocardiographic marker of arrhythmogenesis that reflects the degree of heterogeneity in myocardial repolarization. The TpTe interval, measured as the time from the peak of the T wave to the end of the T wave, and the TpTe/QT ratio, calculated by dividing the TpTe interval by the QT interval, were assessed at baseline (visit 1, day 0) and follow-up (final visit, approximately 90 days later).
  Prolonged TpTe and TpTe/QT intervals are associated with a higher risk of sudden cardiac death (SCD) in various cardiac conditions, including hypertrophic cardiomyopathy and long QT syndrome, making them valuable prognostic markers. In this study, 12-lead ECGs were recorded using Micromed electronic equipment (configured at a paper speed of 25 mm/s and amplitude of 10 mm/mV), and intervals were manually measured with Wincardio software (version 11.1.0.0).
Effect of Dapagliflozin on the J-Tpeak Interval | 90 days
  The J-Tp interval (JTp), an important marker of delays in the early phase of the action potential, was measured from the J point to the peak of the T wave (Tp) on 12-lead electrocardiograms (ECGs). Baseline ECG recordings were conducted at visit 1 (day 0), while follow-up recordings were obtained approximately 90 days later at the final visit.
  All ECGs were recorded using Micromed electronic equipment, standardized with a paper speed of 25 mm/s and an amplitude of 10 mm/mV. Manual measurements of the JTp interval were performed using Wincardio software (version 11.1.0.0). This parameter was assessed to evaluate the effect of dapagliflozin on early ventricular repolarization dynamics, providing valuable insights into potential delays in the initial phase of the cardiac action potential and contributing to the overall understanding of its impact on cardiac electrophysiology.
Effect of Dapagliflozin on the QT interval dispersion (QTd) | 90 days
  QT interval dispersion (QTd), a marker of spatial heterogeneity in ventricular repolarization, was calculated as the difference between the longest (QTmax) and shortest (QTmin) QT intervals measured on 12-lead electrocardiograms (ECGs). Baseline ECG recordings were taken at visit 1 (day 0), and follow-up recordings were acquired approximately 90 days later at the final visit.
  The ECGs were obtained using Micromed electronic equipment, configured with a paper speed of 25 mm/s and an amplitude of 10 mm/mV. All interval measurements were manually conducted using Wincardio software (version 11.1.0.0) to ensure precision and standardization.
  This parameter was analyzed to assess the impact of dapagliflozin on reducing ventricular repolarization dispersion, which has been associated with an increased risk of arrhythmias and sudden cardiac death (SCD) in patients with type 2 diabetes.
Effect of Dapagliflozin on The QRS-T angle | 90 days
  The QRS-T angle, a vectorcardiographic marker of ventricular repolarization heterogeneity and electrical dyssynchrony, was evaluated using data obtained from 12-lead electrocardiograms (ECGs). Baseline ECGs were recorded at visit 1 (day 0), and follow-up recordings were performed approximately 90 days later at the final visit.
  The QRS-T angle was calculated by analyzing the electrical axes of the QRS complex and the T wave in the frontal plane leads. These measurements were performed using the MYEKG software, which processed the R and T wave amplitudes in millimeters and calculated the spatial QRS-T angle using a dedicated algorithm available at [https://pt.my-ekg.com/calculadoras-ecg/calculadora-eixo-eletrico.php].
  The QRS-T angle was categorized into three groups: normal (0 to 105°), borderline (105 to 135°), and abnormal (135 to 180°). This parameter was assessed to determine the impact of dapagliflozin on ventricular electrical heterogeneity
Effect of Dapagliflozin on the Heart rate | 90 days
  Heart rate was measured from 12-lead electrocardiograms (ECGs) recorded during designated outpatient visits. Baseline ECG recordings were obtained at visit 1 (day 0), and follow-up ECGs were performed approximately 90 days later at the final visit.
  The ECGs were recorded using Micromed electronic equipment, standardized with a paper speed of 25 mm/s and an amplitude of 10 mm/mV. Heart rate measurements were automatically calculated by the Wincardio software (version 11.1.0.0) and manually verified when necessary to ensure precision and consistency.
  This parameter was evaluated to assess the effect of dapagliflozin on overall cardiac rhythm and rate regulation in patients with type 2 diabetes. Independent external examiners reviewed all ECGs to ensure objectivity and reliability in the study data.

OTHER OUTCOMES:
Glycated hemoglobin (HbA1c) | 90 days
  The measurement of glycated hemoglobin (HbA1c %) was performed through venous blood collection, with samples sent for analysis in a certified laboratory in accordance with the international quality standards established by the National Glycohemoglobin Standardization Program (NGSP) and aligned with the reference methods of the International Federation of Clinical Chemistry (IFCC).
  The collected data were recorded in the study's digital Case Report Form (CRF) during the baseline visit and again after 90 days, at the end-of-study visit.
Weight | 90 days
  he participants' weight (Kg) was measured using a properly calibrated scale, with participants standing upright, barefoot, and wearing light clothing. The data were recorded in the study's digital Case Report Form (CRF) during the baseline visit and again after 90 days, at the end-of-study visit, to monitor any changes associated with the treatment or clinical progression.
Body Mass Index (BMI) | 90 days
  The participants' Body Mass Index (BMI) was calculated using the formula weight (kg) divided by height squared (m²), based on measurements obtained during the baseline visit. Weight was measured using a properly calibrated scale, and height was measured with a stadiometer, with participants standing barefoot and in an upright position. The BMI data were recorded in the study's digital Case Report Form (CRF) during the baseline visit and again after 90 days, at the end-of-study visit, to assess any changes associated with the treatment or clinical progression.
Systolic and Diastolic Blood Pressure | 90 days
  The participants' systolic and diastolic blood pressure (BP) was measured in millimeters of mercury (mmHg) using a properly calibrated automated or manual sphygmomanometer. Measurements were taken with participants seated, at rest for at least five minutes, and with their arm supported at heart level. Blood pressure readings were recorded in triplicate, with the average value documented for accuracy.
  The systolic and diastolic BP data were entered into the study's digital Case Report Form (CRF) during the baseline visit and again after 90 days, at the end-of-study visit, to monitor any changes associated with the treatment or clinical progression.
Glomerular Filtration Rate | 90 days
  The participants' glomerular filtration rate (GFR) was estimated in milliliters per minute per 1.73 square meters (mL/min/1.73 m²) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. This calculation was based on serum creatinine levels, age, sex, and race, obtained from blood samples analyzed in a certified laboratory.
  The GFR data were recorded in the study's digital Case Report Form (CRF) during the baseline visit and again after 90 days, at the end-of-study visit, to evaluate renal function changes associated with the treatment or clinical progression.
Echocardiographic - Left ventricular ejection fraction (LVEF), | 90 days
  The echocardiographic parameter left ventricular ejection fraction (LVEF), expressed as a percentage (%), was evaluated using standard transthoracic echocardiography (TTE).
  All measurements were conducted by certified sonographers using clinically approved equipment, adhering to the guidelines established by the American Society of Echocardiography (ASE). Data collected during the echocardiographic assessments were systematically documented in the study's digital Case Report Form (CRF). Evaluations were performed both at the baseline visit and at the end-of-study visit (90 days) to monitor potential structural or functional cardiac changes related to the treatment or clinical progression.
Echocardiographic - Left ventricular end-diastolic diameter (LVEDD) | 90 days
  The echocardiographic parameter left ventricular end-diastolic diameter (LVEDD), measured in millimeters (mm), was evaluated using standard transthoracic echocardiography (TTE).
  All measurements were performed by certified sonographers using clinically validated equipment, in compliance with the guidelines of the American Society of Echocardiography (ASE). The obtained echocardiographic data were systematically recorded in the study's digital Case Report Form (CRF). Assessments were conducted at the baseline visit and at the end-of-study visit (90 days) to track any structural cardiac changes associated with treatment or clinical progression.
Echocardiographic - Left ventricular systolic diameter (LVSD) | 90 days
  The echocardiographic parameter left ventricular systolic diameter (LVSD), measured in millimeters (mm), was assessed using standard transthoracic echocardiography (TTE).
  All measurements were performed by certified sonographers utilizing clinically validated equipment, in accordance with the guidelines of the American Society of Echocardiography (ASE). The recorded data were systematically entered into the study's digital Case Report Form (CRF). Measurements were obtained at both the baseline visit and the end-of-study visit (90 days) to evaluate potential changes in ventricular dimensions associated with treatment or clinical progression.
Echocardiographic - Left atrial diameter (LAD) | 90 days
  The echocardiographic parameter left atrial diameter (LAD), measured in millimeters (mm), was assessed using standard transthoracic echocardiography (TTE).
  All measurements were performed by trained and certified sonographers utilizing clinically validated equipment, in accordance with guidelines provided by the American Society of Echocardiography (ASE). The collected LAD data were systematically recorded in the study's digital Case Report Form (CRF) during the baseline visit and again at the end-of-study visit (90 days) to evaluate potential changes in left atrial size associated with treatment effects or clinical progression.
Key Medications in Use | 90 days
  The use of key medications, including beta-blockers, propafenone, amiodarone, renin-angiotensin-aldosterone system inhibitors (RAAS inhibitors), angiotensin II receptor blockers (ARBs), sacubitril-valsartan, and mineralocorticoid receptor antagonists (MRAs), was documented for each participant. Information on medication type, dose, and frequency was collected during interviews and confirmed through medical records.
  These data were systematically recorded in the study's digital Case Report Form (CRF) during the baseline visit and again after 90 days, at the end-of-study visit, to monitor ongoing treatment regimens and assess their potential influence on clinical outcomes.
Hospitalization Within 90 Days | 90 days
  The variable for hospitalization within 90 days was recorded as a categorical variable (Yes/No). These data were collected during the final visit at 90 days, based on self-reported information provided by the participant or through active data retrieval from medical records and hospital databases to ensure accuracy.
  The hospitalization data were documented in the study's digital Case Report Form (CRF) during the 90-day visit to assess the occurrence of hospital admissions during the study period and their potential influence on outcomes.
All-Cause Mortality | 90 days
  The variable for all-cause mortality was recorded as a categorical variable (Yes/No). These data were collected during the final visit at 90 days through direct communication with the participant's family or caregiver, or via active data retrieval from medical records, hospital databases, or public death registries to ensure accuracy.
  The all-cause mortality data were documented in the study's digital Case Report Form (CRF) at the 90-day visit to assess the occurrence of death from any cause during the study period and its potential impact on clinical outcomes.
Cause of Death (Cardiovascular or Non-Cardiovascular) | 90 days
  The cause of death was recorded as a categorical variable, classified as either cardiovascular death or non-cardiovascular death. These data were collected during the final visit at 90 days through direct communication with the participant's family or caregiver, or via active data retrieval from medical records, hospital databases, or public death registries. For cardiovascular deaths, the classification was based on standard clinical definitions, including sudden cardiac death, death due to myocardial infarction, stroke, or other cardiovascular causes.
  The cause-of-death data were documented in the study's digital Case Report Form (CRF) at the 90-day visit to differentiate between cardiovascular and non-cardiovascular mortality and to assess its potential influence on clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital Beneficencia Portuguesa de São Paulo, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campos RN, Moreira DAR, Fonseca GM. Effect of dapagliflozin, a sodium-glucose co-transporter 2 inhibitor, on ventricular repolarization electrocardiographic parameters in type 2 diabetes patients: DAPA - ECG study. Front Clin Diabetes Healthc. 2025 Mar 31;6:1537005. doi: 10.3389/fcdhc.2025.1537005. eCollection 2025. PMID 40230406